CLINICAL TRIAL: NCT06523972
Title: Promoting Cardiovascular Disease Awareness and Cardiovascular Health Among Minnesota State Fair Attendees: The Great Minnesota Heart Health Check
Brief Title: A Study of Cardiovascular Disease Awareness and Cardiovascular Health
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Principal Investigator, Mayo Clinic
Other Study IDs: 24-006211
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Diseases; Cardiovascular Health
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective is to increase awareness of various cardiovascular diseases (CVDs) through an interactive, educational experience to promote cardiovascular health (CVH) via an inflatable heart model exhibit and assess community CVD knowledge and whether this experience is an acceptable tool to promote and provide education on CVH.

ELIGIBILITY:
Inclusion Criteria:

* MN resident
* Active email address
* ≥18 years of age

Exclusion Criteria:

- Inability to speak, read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years of age)
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Health (CVH) | Baseline
  CVH will be measured by LE8 composite score (scale 0-100 points). A higher composite score is associated with ideal cardiovascular health.

SECONDARY OUTCOMES:
Social Determinants of Health (SDoH) | Baseline
  SDoH will be measured by education level, insurance status, and neighborhood zip code
Individual LE8 component scores (Life's Essential 8) | Baseline
  LE8 component scores will be measured from eight health behavior and clinical factors including diet, physical activity, nicotine exposure, sleep health, body mass index (BMI), blood lipids, blood pressure (BP), and blood glucose.

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess Brewer, M.D., M.P.H., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States